CLINICAL TRIAL: NCT06586151
Title: Harnessing the Power of Technology to Develop a Population-based HIV Prevention Program for Trans Girls
Brief Title: Testing a Gender-inclusive HIV Prevention Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: University of Miami (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01NR020309 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: HIV Prevention
Keywords: HIV; Adolescence; mHealth

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants, but not researchers, will be blinded to study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information, Motivation and Skills arm (Experimental): Text messaging-based program that lasts 5 months. Content includes information, motivation and behavioral skills about how to prevent HIV, as well as information about healthy and unhealthy romantic relationships, and navigating issues related to one's gender.
  Interventions: Behavioral: Transcendent Health
- Information Only arm (Placebo Comparator): Text messaging-based program that lasts 5 months. Content includes information about HIV prevention and aspects of a healthy adolescent lifestyle (e.g., self-esteem).
  Interventions: Behavioral: Text Messaging with Information

INTERVENTIONS:
Behavioral: Transcendent Health — Gender-inclusive HIV prevention program: Text messaging-based program that lasts 5 months. Content includes information, motivation and behavioral skills about how to prevent HIV, as well as information about healthy and unhealthy romantic relationships, and navigating issues related to one's gender.
  Arms: Information, Motivation and Skills arm
Behavioral: Text Messaging with Information — Text messaging-based program that lasts 5 months. Content includes information about HIV prevention and aspects of a healthy adolescent lifestyle (e.g., self-esteem).
  Arms: Information Only arm

SUMMARY:
If, over time, data suggest the intervention impacts HIV preventive behavior at the population level, it will be unique in that it can be quickly and cost effectively scaled up to impact thousands of trans girls and nonbinary youth assigned male at birth.

ELIGIBILITY:
Inclusion Criteria:

1. assigned male sex at birth and currently have a non-cisgender identity (e.g., transgender girl, non-binary, gender fluid, unsure);
2. aged 14-18 years and have not yet graduated high school;
3. English-speaking;
4. the sole user of a cell phone with an unlimited text messaging plan;
5. have access to the Internet to complete online surveys;
6. intend to have the same cell number for the next 6 months;
7. provide informed assent;
8. not have taken part in a previous #TranscendentHealth study activity or know someone who is in the study to increase the diversity of input from transgirls, and
9. agree to enroll over the phone with study staff.

Exclusion Criteria:

* None beyond not meeting inclusion criteria

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Transgender girls and non-binary youth; not exclusively cisgender identified
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number testing for HIV and/or sexual transmitted infections | At any time after baseline through 8-months.
  Self report of having been tested for either HIV or a sexually transmitted infection

SECONDARY OUTCOMES:
Number Taking PreExposure Prophylaxis (PrEP) for HIV | At any time after baseline through 8-months.
  Self-report of taking PrEP at any time since the prior assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovative Public Health Research, San Clemente, California, United States

IPD SHARING:
Plan to Share IPD: No